CLINICAL TRIAL: NCT06719388
Title: Exercise Therapy Combined with a Jaw-Mobilizing Device for Improving Maximal Mouth Opening and Trismus in Patients with Head and Neck Cancer: a Randomized Controlled Trial
Brief Title: Exercise Therapy and Jaw-Mobilizing Device for Trismus in Head and Neck Cancer Patients
Acronym: ET-JMD for Tri
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Tsai-Wei Huang, Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Jaw-Mobilizing Device
Record Dates: First submitted 2024-11-28; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Head and Neck Cancers; Trismus; Radiotherapy Side Effects
Keywords: Head and Neck Cancer; Trismus; Radiotherapy-Induced Mouth Opening Limitation
MeSH Terms: conditions — Head and Neck Neoplasms; Trismus

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two parallel groups: the experimental group, which receives exercise therapy combined with a jaw-mobilizing device, or the control group, which receives exercise therapy only. Both groups are followed concurrently throughout the study period.
Who Masked: Participant
Masking Description: Participants are unaware of their group allocation (experimental or control) to minimize bias in self-reported outcomes and adherence to the intervention. However, investigators and outcome assessors are not masked due to the nature of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Participants in the experimental group will receive a combination of exercise therapy and a jaw-mobilizing device. The intervention includes structured exercise therapy sessions and the use of the jaw-mobilizing device for 12 weeks, beginning one week prior to radiotherapy. Follow-ups will occur at weeks 16, 24, and 36 to assess outcomes.
  Interventions: Behavioral: combination of exercise therapy and a jaw-mobilizing device
- Control Group (Placebo Comparator): Participants in the control group will receive exercise therapy only. This intervention involves the same structured exercise therapy sessions as the experimental group for 12 weeks, beginning one week prior to radiotherapy. Follow-ups will occur at weeks 16, 24, and 36 to assess outcomes.
  Interventions: Behavioral: exercise therapy only

INTERVENTIONS:
Behavioral: combination of exercise therapy and a jaw-mobilizing device — Participants in the experimental group will receive a combination of exercise therapy and a jaw-mobilizing device. The intervention includes structured exercise therapy sessions and the use of the jaw-mobilizing device for 12 weeks, beginning one week prior to radiotherapy. Follow-ups will occur at weeks 16, 24, and 36 to assess outcomes.
  Arms: Experimental Group
Behavioral: exercise therapy only — Participants in the control group will receive exercise therapy only. This intervention involves the same structured exercise therapy sessions as the experimental group for 12 weeks, beginning one week prior to radiotherapy. Follow-ups will occur at weeks 16, 24, and 36 to assess outcomes.
  Arms: Control Group

SUMMARY:
This study evaluates the effects of exercise therapy combined with a jaw-mobilizing device on enhancing quality of life in head and neck cancer patients undergoing radiotherapy.

DETAILED DESCRIPTION:
This study investigates the efficacy of exercise therapy combined with a jaw-mobilizing device (ET-JMD) in improving maximal mouth opening (MMO), preventing trismus, enhancing quality of life (QoL), and alleviating trismus-related symptoms in head and neck cancer (HNC) patients undergoing radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years.
* Ability to communicate in Mandarin or Taiwanese, without significant reading, hearing, or writing impairments, and capable of completing questionnaires independently or with researcher assistance.
* Diagnosed with head and neck cancer and scheduled for initial radiotherapy to the head and neck region.
* Clear consciousness without severe cognitive or psychiatric disorders.
* Presence of intact central incisors (#11, #41) on the right side or (#21, #31) on the left side of both the upper and lower jaws.
* Baseline maximal mouth opening (MMO) ≥ 25 mm.
* Willingness to participate in the study with signed informed consent.

Exclusion Criteria:

* Known temporomandibular joint disorders.
* Postoperative wound healing complications diagnosed by a physician that prevent participation in mouth-opening rehabilitation exercises.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Maximal Mouth Opening | Baseline to Week 36
  Change in Maximal Mouth Opening (MMO) from Baseline to Week 36. higher score means worse.

SECONDARY OUTCOMES:
Quality of Life Scores | Baseline to Week 36
  Change in Quality of Life Scores (EORTC QLQ-H&N35) from Baseline to Week 36. higher score means good quality.
Trismus-Related Symptom Distress Scores | Baseline to Week 36
  Change in Trismus-Related Symptom Distress Scores (GTQ2) from Baseline to Week 36. higher score means worse.

CONTACTS AND LOCATIONS:
Locations (1):
- tri-Service Gereral Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol